CLINICAL TRIAL: NCT01673568
Title: Postoperative Abdominal Binder in Reducing Seroma Formation and Pain After Ventral (Umbi/Epi) Hernia Repair.
Brief Title: Abdominal Binder to Reduce Pain and Seroma Formation
Acronym: ABD- BINDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Mette Willaume Christoffersen, MD, PhD. stud., Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AB-BINDER
Record Dates: First submitted 2012-07-04; First posted 2012-08-28 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Ventral Hernias
MeSH Terms: conditions — Hernia, Ventral | interventions — Trusses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- abdominal binder (Active Comparator): The abdominal binder is worn from immediately after the operation and continuously for 7 days, night and day. The belts are standard elastic belts (ostomy belts) from "ETO garments©" with standard height of 22 cm. and five different sizes in width (S, M, L, XL, XXL- depending on waist measure). A fitting will be done before the operation by waist measurement according to the recommendation from the company.
  Interventions: Device: ETO garments
- no abdominal binder (No Intervention): no abdominal binder

INTERVENTIONS:
Device: ETO garments — patients wearing abdominal binder for 7 days postoperatively
  Other Names: longuette; ostomy belt; trusses; girdle
  Arms: abdominal binder

SUMMARY:
Postoperative seroma formation is one of the most common complications after ventral hernia repair. Although some seromas may not have clinical impact, postoperative seroma formation often causes pain and discomfort and may even compromise wound healing. The use of postoperative abdominal binder is often recommended after ventral hernia repair to prevent seroma and diminish pain, but still with no scientific evidence. The primary aim of the present study is to investigate the effect of postoperative abdominal binders after laparoscopic ventral hernia repair on postoperative pain, discomfort and quality of life. Secondary, we register seroma formation.

Method and material Randomized, controlled, multi-center, investigator-blinded study. A minimum of 56 patients (2X28 umbi/epi) are included, inclusion number is based on power calculations. Patients are randomized either to abdominal binder or no abdominal binder. The abdominal binder is worn from immediately after the operation and continuously for 7 days, night and day. Outcomes are based on patient self-reported registrations using Visual Analog Scales (VAS) and Carolina Comfort Scale (CCS), which is a validated, hernia-specific tool to estimate quality of life, pain and discomfort. Patients are followed-up for 30 days. For secondary outcome we use ultrasound to measure the volume of seroma formation. We use Mann-Witney, non-parametric statistics calculating the seroma formation and Friedmanns test for pain, discomfort and quality of life for the effect of time on inter- and intragroup differences during the study period. P < 0.05 is considered significant.

DETAILED DESCRIPTION:
Postoperative seroma formation is one of the most common complications after ventral hernia repair. Although some seromas may not have clinical impact postoperative seroma formation often causes pain and discomfort and may even compromise wound healing. Several interventional procedures have been investigated to reduce or avoid postoperative seroma formation such as removal of the hernia sac, VAC (vacuum-assisted closure) therapy, talcum application to the subcutaneous layer, suction etc., but results are conflicting and evidence is of poor quality. The use of postoperative abdominal binder is often recommended after ventral hernia repair to prevent seroma and diminish pain, but still with no scientific evidence. Randomized, controlled, multi-center, investigator-blinded study supplemented with blinded statistical analysis (see below). 56 patients (2 x 28, umbi/epi) Due to power calculations. An intention to treat analysis is done. Patients are randomized either to abdominal binder or no abdominal binder. The abdominal binder is worn from immediately after the operation and continuously for 7 days, night and day. The belts are standard elastic belts (ostomy belts) from "ETO garments©" with standard height of 22 cm. and five different sizes in width (S, M, L, XL, XXL- depending on waist measure). A fitting will be done before the operation by waist measurement according to the recommendation from the company. Patients are followed-up for 30 days with clinical follow-up at day 7 and 30.

ELIGIBILITY:
Inclusion Criteria:

* Elective, primary and recurrent laparoscopic umbilical and epigastric hernia repair with mesh reinforcement
* Fascia defects 2-8 cm measured preoperatively by the surgeon at the out-patient clinic for umbi/epi
* Elective, primary and recurrent laparoscopic trocar-site hernia
* Patients between 18-80 years

Exclusion Criteria:

* Open ventral hernia repair
* Expected low compliance (language problems, dementia and abuse etc.)
* Fascia defects >8 cm at the preoperative clinical examination.
* Acute operation
* Chronic pain syndrome
* Decompensated liver cirrhosis (Child-Pugh B-C)
* Patients with a stoma
* If a secondary operation is performed during the hernia repair procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thue Bisgaard, MD, Study Director — University Hospital HVidovre
Locations (1):
- Hvidovre Hospital, Hvidovre, CPH, Denmark

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abdominal Binder | no Abdominal Binder
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: patiens were median 51 years, gender M:F=22:6.
Groups:
- no Abdominal Binder: no abdominal binder was warn
- Total: Total of all reporting groups
Arm/Group | Abdominal Binder | no Abdominal Binder | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Median (Full Range); unit: years] | 51 [21 to 73] | 51 [31 to 71] | 51 [21 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale of Pain Activity
Description: Outcome is based on patient self-reported registrations using Visual Analog Scales (VAS) where 0 is no pain in activity and 100 is worst imaginable pain in activity.
Time Frame: 24 hours after hernia repair
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Abdominal Binder | no Abdominal Binder
Number analyzed (Participants) | 28 | 28
units on a scale | 50 [13 to 100] | 70 [11 to 97]

2. Secondary Outcome: Seroma Formation
Description: Seroma formation measured on day 7 postoperatively with trans abdominal ultrasound scan (US). The method used in this study to estimate the volume of seroma is to measure the longitudinal section and cross section of the effusion and thereby calculating the volume.
Time Frame: postoperative day 7
Measure: Median (Full Range); unit: mL
Arm/Group | Abdominal Binder | no Abdominal Binder
Number analyzed (Participants) | 28 | 28
mL | 7 [0 to 300] | 9 [0 to 163]

ADVERSE EVENTS:
Arm/Group | Abdominal Binder | no Abdominal Binder
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No